CLINICAL TRIAL: NCT07339228
Title: Meet Me on the Pitch: Developing and Testing a Community-Based Sports and Behavioral Health Intervention for Youth
Acronym: MMotP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Soccer Without Borders (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A144370; U01NR021576 (NIH)
Record Dates: First submitted 2026-01-12; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Mental Health; Psychological Well Being; Adolescent Health; Help-Seeking Behavior
Keywords: Adolescent; Behavioral health; Well-being; Sports; School engagement; Social connection
MeSH Terms: conditions — Psychological Well-Being; Help-Seeking Behavior

STUDY DESIGN:
Intervention Model Description: Participants are individually randomized within soccer teams to either the intervention group (MMotP program + Soccer Without Borders standard programming) or the control group (standard Soccer Without Borders programming only). MMotP consists of six one-hour sessions delivered weekly.
Who Masked: Outcomes Assessor
Masking Description: The youth participants and coaches enrolling participants will not know of study assignment until after completing recruitment, consent and the baseline survey. At that point, the UCSF study team will use a random number generator to assign each participant to the intervention or control condition. The researcher conducting the outcomes analysis will not know the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Standard Programming) (No Intervention): Participants will continue regular Soccer Without Borders programming, including soccer practices and team-building activities with their coach.
- Intervention Group (MMotP Program + Standard Programming) (Experimental): In addition to standard Soccer Without Borders programming, participants will receive MMotP, a six-session behavioral health intervention. MMotP sessions will be delivered weekly by their trained coach outside of soccer practices.
  Interventions: Behavioral: Meet Me on the Pitch (MMotP)

INTERVENTIONS:
Behavioral: Meet Me on the Pitch (MMotP) — Meet Me on the Pitch is a six-session behavioral health intervention delivered by trained Soccer Without Borders coaches to small groups of youth, ages 14-21. Sessions are held weekly at school sites, typically after school. The six one-hour sessions follow a consistent structure that includes a brief preview of the day's session and a review of the prior session; three learning goals; and worksheets and play-based activities to facilitate learning and reinforce key concepts. In Session 1, participants explore identities and identify values to help guide action in future sessions. In Session 2, participants establish a personal or academic goal, identify barriers and facilitators, and set an actionable step to support their goal by the following session. In Session 3, coaches introduce the DNA-V model and help participants develop psychological skills to reach their goals. In Session 4- 6, participants use the DNA-V Discussion Tool and plan additional short-term actionable steps to con
  Arms: Intervention Group (MMotP Program + Standard Programming)

SUMMARY:
This study evaluates Meet Me on the Pitch (MMotP), a community-based intervention that integrates sports, schools, and behavioral health with the goal of improving the behavioral health, well-being and academic performance of youth. MMotP is a novel approach that builds on evidence-based practices by using sports as a means to foster social-emotional development and address barriers to academic, health, and social services. The study assesses feasibility, acceptability, and short-term outcomes through a randomized controlled trial comparing MMotP to standard sports programming. The intervention will be implemented by the non-profit organization Soccer Without Borders and evaluated by the University of California, San Francisco.

DETAILED DESCRIPTION:
Meet Me on the Pitch (MMotP) is an innovative community-based intervention designed to improve the behavioral health, well-being and academic performance of youth (ages 14-21). The six-session intervention combines soccer-based activities with behavioral health education using the DNA-V model, a youth-focused adaptation of Acceptance and Commitment Therapy (ACT). By training trusted community members, specifically soccer coaches, to deliver a tailored behavioral health intervention, MMotP addresses barriers to academic, health, and social services while fostering social-emotional development.

This study evaluates MMotP through a parallel randomized controlled trial. Youth participants will be randomized within their soccer teams to either the supplemental MMotP intervention or just standard sports programming. The study will assess changes in primary outcomes, including mental health (psychological flexibility and self-efficacy) and academic support-seeking behaviors, as well as secondary outcomes related to social connection, school engagement, and access to services. Youth will complete surveys at baseline, 3 months, and 6 months to measure these outcomes.

MMotP will be implemented by Soccer Without Borders in the San Francisco Bay Area and Colorado and evaluated by the University of California, San Francisco. This study is funded by the National Institute of Nursing Research.

ELIGIBILITY:
Inclusion Criteria:

* Youth ages 14-21 participating in Soccer Without Borders programming
* Regular attendance at team soccer practice
* Ability to speak English or Spanish

Exclusion Criteria:

* Youth who do not participate in Soccer Without Borders activities
* Youth who do not attend soccer practice regularly
* Youth who do not speak English or Spanish
* Youth who have already received the MMotP program

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 480 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychological Flexibility | Baseline, 3-month follow-up, 6-month follow-up
  Self-reported response to the Avoidance & Fusion Questionnaire (AFQ-Y8), using 8-item version adapted for youth. Each item is scored on a 4-point Likert scale from 1 (Not at All True) to 4 (Very Much True). Responses are summed for a total score.
Self-Efficacy | Baseline, 3-month follow-up, 6-month follow-up
  Self-reported response to the General Self-Efficacy Scale (GSE), using 10-item version adapted for youth. Each item is scored on a 5-point Likert scale from 1 (Never) to 5 (Very Often). Responses are summed for a total score.
Help-seeking for Academic Needs | Baseline, 3-month follow-up, 6-month follow-up
  Self-reported response to four UCSF-developed items: awareness of adult at school for academic support (Yes/No/Not Sure), need for academic support in past month (Yes/No/Not Sure), sought academic support in past month (Yes/No), and willingness to seek academic support in future (Definitely No/Probably No/Probably Yes/Definitely Yes).

SECONDARY OUTCOMES:
Social Connection | Baseline, 3-month follow-up, 6-month follow-up
  Self-reported response to California Healthy Kids Survey (CHKS) Co-Regulation Supports Scale (Home Adult and Peer) and Community Supports Scale. Each item is scored on a 4-point Likert scale from 1 (Not at All True) to 4 (Very Much True). Responses are average for a mean score.
School Engagement | Baseline, 3-month follow-up, 6-month follow-up
  Self-reported school attendance in the past month. Self-reported recent academic grades. Self-reported response to California Healthy Kids Survey (CHKS) Internal Assets - Educational Goals Scale. Each item is scored on a 4-point Likert scale from 1 (Not at All True) to 4 (Very Much True). Responses are average for a mean score.
Help-seeking for Health and Social Service Needs | Baseline, 3-month follow-up, 6-month follow-up
  Self-reported response to UCSF-developed items: awareness of support (Yes/No/Not Sure), need for support in past month (Yes/No/Not Sure), sought support in past month (Yes/No), and willingness to seek support in future (Definitely No/Probably No/Probably Yes/Definitely Yes).

CONTACTS AND LOCATIONS:
Overall Officials: Mara Decker, DrPH, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Soccer Without Borders - Bay Area, Oakland, California
  - Soccer Without Borders - Colorado, Denver, Colorado

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant survey data will be made available for secondary analyses. Given the study's focus on a particularly vulnerable population (i.e., minors), we limit data sharing to scientists approved by the UCSF research team and Institutional Review Board. Because of the nature of the data and potential risks to research participants, our datasets will not be placed in a data repository. Data will be shared in compliance with UCSF IRB-approved protocols and NIH data-sharing requirements.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available on or before December 2029.
Access Criteria: Sharing access criteria are under development.